CLINICAL TRIAL: NCT06909929
Title: Pemberian Lipid Intravena Dosis Tinggi Untuk Bayi Sangat Prematur Atau Berat Lahir Sangat Rendah Terhadap Pertumbuhan
Brief Title: High-Dose Intravenous Lipid for Very Preterm or Very Low Birth Weight Infants Effects on Growth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Putri Maharani Tristanita Marsubrin, MD, PhD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LIPIP2GVS1G
Record Dates: First submitted 2024-12-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Very Preterm Birth
MeSH Terms: interventions — Lipid IV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2 gram (Experimental): This group will get 2 g of lipid IV in the early 24 hours of life
  Interventions: Dietary Supplement: Lipid IV 2 g
- 1 gram (Active Comparator): This group will get 1 g of lipid IV in the early 24 hours of life
  Interventions: Dietary Supplement: lipid IV 1 gram

INTERVENTIONS:
Dietary Supplement: Lipid IV 2 g — This group will get 2 g of lipid IV in the early 24 hours of life
  Arms: 2 gram
Dietary Supplement: lipid IV 1 gram — This group will get 1 g of lipid IV in the early 24 hours of life
  Arms: 1 gram

SUMMARY:
This is a RCT study conducted in Cipto Mangunkusumo Hospital in very preterm infants. The investigators compared early intravena lipid start with 2 gram per body weight and 1 gram per body weight and observed the time to reach birth weight.

DETAILED DESCRIPTION:
Neonates with <32 weeks gestation age or <1500 gram birth weight gets early intravena lipid start with 2 gram per body weight and 1 gram per body weigh then observed the time to reach birth weight

ELIGIBILITY:
Inclusion Criteria:

* birth weight below 1500 gram or gestational age below 32 weeks

Exclusion Criteria:

* mayor congenital abnormalities

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
return to birth weight | day
  time of the participants to reach back the birth weight up to 28 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Putri MT Marsubrin, MD, PhD, Principal Investigator — Cipto Mangunkusumo Hospital, Jakarta, Central Jakarta 10430
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Central Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No